CLINICAL TRIAL: NCT07090759
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase III Trial of GST-HG141（Neracorvir）for Combination Therapy (add-on) in Patients With Inadequate Response to Antiviral Drugs in Chronic Hepatitis B (CHB)
Brief Title: To Evaluate the Efficacy, Safety and Population Pharmacokinetics of GST-HG141 in Patients With Chronic Hepatitis B (CHB) Who Have an Inadequate Response to Antiviral Drug Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GST-HG141-III-01
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GST-HG141 (Experimental)
  Interventions: Drug: GST-HG141
- GST-HG141 Placebo (Placebo Comparator)
  Interventions: Drug: GST-HG141 Placebo

INTERVENTIONS:
Drug: GST-HG141 — GST-HG141 50 mg BID
  Arms: GST-HG141
Drug: GST-HG141 Placebo — GST-HG141 Placebo BID
  Arms: GST-HG141 Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial, aiming to evaluate the efficacy and safety of GST-HG141 in patients with chronic hepatitis B who have an inadequate response to antiviral drug treatment.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial, aiming to evaluate the efficacy and safety of GST-HG141 in patients with chronic hepatitis B who have an inadequate response to antiviral drug treatment.

This research project enrolled a total of 526 CHB patients who have an inadequate response to hepatitis B antiviral treatment. They were divided into two groups, with 263 patients in each group.

The qualified participants were randomly assigned to the GST-HG141 group and the placebo group at a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals aged 18-70 years (inclusive of the boundaries);
2. Male weight ≥ 50 kg, female weight ≥ 45 kg, with a body mass index (BMI) within the range of 18-35 kg/m2 (inclusive of the boundaries);
3. Have been continuously taking nucleoside analogues (entecavir [ETV], tenofovir disoproxil fumarate [TDF], emivirofavir [TMF], or propivirofavir [TAF]) for more than one year (with a break of less than one month in the past year), and are receiving treatment at the time of screening and agree to accept the treatment plan provided by this study during the study period;

   * Have maintained the same NA monotherapy for more than 3 months before screening
4. HBeAg positive, serum HBV DNA can be detected by high-sensitivity PCR, and HBV DNA > 50 IU/mL;
5. At the time of screening, ALT ≤ 5×ULN;
6. Male participants with a fertile female partner or female participants of childbearing age who are willing to voluntarily take effective contraceptive measures from the time of screening until 28 days after the completion of the study ;
7. Sign the informed consent form before the trial and be able to complete the study as required by the trial protocol.

Exclusion Criteria:

1. History of life-threatening severe allergic reactions such as anaphylactic shock, or allergy to the active ingredients or excipients of the study drug as suspected by the investigator;
2. Concomitant use of cytochrome P450 enzyme 3A4 (CYP3A4) inhibitors, inducers, or substrates within 28 days prior to screening;
3. Systemic use of immunosuppressants, immunomodulators (interferon must be discontinued for more than 12 months), or cytotoxic drugs within 6 months prior to screening; or vaccination with live attenuated vaccines within 1 month prior to screening;
4. Presence of acute infections requiring treatment prior to randomization;
5. Clinically significant acute or chronic liver disease not caused by HBV infection, rendering the subject unsuitable for participating in the study as determined by the investigator;
6. Subjects with a history of cirrhosis (e.g., subjects who have undergone pathological examination of liver tissue with a report indicating cirrhosis or those who have undergone endoscopy indicating esophageal or gastric varices); or subjects with currently diagnosed or suspected decompensated cirrhosis, including but not limited to: hepatic encephalopathy, hepatorenal syndrome, bleeding from esophageal or gastric varices, splenomegaly, and ascites; or subjects with significant progression of liver fibrosis;
7. Primary liver cancer; serum alpha-fetoprotein (AFP) greater than 20 μg/L (or 20 ng/mL) or DCP>40 mAU/mL or imaging suggesting possible malignant lesions in the liver; concurrent other malignancies or history of other malignancies within the past 5 years (except for cured basal cell carcinoma or squamous cell carcinoma of the skin and cervical carcinoma in situ);
8. Presence of gastrointestinal impairment or gastrointestinal disease that may affect the absorption of oral medication in the judgment of the investigator, such as severe gastrointestinal diseases (peptic ulcer, erosive or atrophic gastritis), partial gastrectomy, Grade > 2 gastrointestinal symptoms at screening (e.g., nausea, vomiting, or diarrhea), etc.;
9. Concurrent severe diseases of the circulatory, respiratory, urinary, hematologic, metabolic, immune, psychiatric, neurological, renal, or other systems, rendering the subject unsuitable for participating in the study as determined by the investigator.
10. Subjects with major trauma or major surgery within 3 months prior to screening; or those who plan to undergo surgery during the study period;
11. Laboratory tests:

    1. Platelet count < 100 × 109/L;
    2. White blood cell count < 3.0 × 109/L;
    3. Absolute neutrophil count < 1.3 × 109/L;
    4. Serum total bilirubin > 2× ULN;
    5. Albumin < 35 g/L;
    6. GFR ≤ 60 mL·min-1·(1.73 m2)-1 (calculated using the CKD-EPI formula);
    7. International normalized ratio (INR) of prothrombin time >1.5;
12. Positive for hepatitis C antibody, positive for HIV antigen/antibody, or positive for syphilis antibody with a positive RPR or TRUST test result;
13. History of sustained alcohol abuse within the past 3 years (weekly alcohol intake > 14 units, where 1 unit of alcohol equals 1 bottle of 350 mL beer, 120 mL wine, or 30 mL of spirits at 40% alcohol content);
14. History of drug dependence or substance abuse;
15. Participation in clinical trials involving other investigational drugs or medical devices and receiving the investigational drug or using the medical device within 3 months prior to screening;
16. Women who are breastfeeding or tested positive for pregnancy;
17. Determined by the investigator to be unsuitable for this trial for any other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with serum Hepatitis B Virus (HBV) DNA | Up to 48 weeks
  Proportion of participants with serum Hepatitis B Virus (HBV) DNA < lower limit of quantification (LLOQ) treatment period;

SECONDARY OUTCOMES:
Serum HBV DNA | Up to 48 weeks
  The changes of HBV DNA level compared to baseline;

CONTACTS AND LOCATIONS:
Locations (1):
- Shulan(Hangzhou) Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No